CLINICAL TRIAL: NCT02604420
Title: Identification of the Pathogenesis of Thrombotic Microangiopathy in the Allo Stem Cell Transplant Setting in Adults
Brief Title: Identification and Treatment of Thrombotic Microangiopathies in Allogeneic Stem Cell Transplants
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1403014892
Record Dates: First submitted 2015-10-15; First posted 2015-11-13 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Thrombotic Microangiopathy; Disorder Related to Bone Marrow Transplantation
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — eculizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells Plasma Bone marrow core biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transplant, no TMA: Adult patients who undergo an allogeneic hematopoietic stem cell transplant but do not meet the criteria for a thrombotic microangiopathy in the one year follow up period. No interventions anticipated.
- Transplant, +TMA: Adult patients who undergo an allogeneic hematopoietic stem cell transplant and meet the criteria for a thrombotic microangiopathy in the one year follow up period. Possible interventions include observation, treatment of an underlying infection or GvHD, use of plasma exchange, or use of anti-complement therapy (eculizumab or other anti-complement drug). Eculizumab is used as a 900mg intravenous infusion over 35 minutes, given weekly for 4 weeks, then 1200mg every other week. Patients must be vaccinated against meningococcus 2 weeks before starting drug or, if that is not feasible because of the physician's assessment of the severity of the TMA, given prophylactic antibiotics for the 2 week period before immunization has taken hold.
  Interventions: Drug: eculizumab

INTERVENTIONS:
Drug: eculizumab
  Other Names: Soliris
  Groups: Transplant, +TMA

SUMMARY:
Mortality in the major thrombotic microangiopathies (TMAs), TTP and aHUS, exceeds 90% unless rapidly diagnosed and appropriately treated. TMAs complicate 10-20% of allogeneic bone marrow hematopoietic stem cell transplants (alloHSCT), conveying inferior survival. Multiple etiologies have been proposed for these transplant-associated TMAs (TA-TMAs), but once infection, graft vs. host disease (GvHD), and drug effects have been ruled out, most are treated as TTP-like disorders using plasma exchange (PEx). But PEx has no impact on mortality in this setting. Clear definition of the pathophysiology of the TA-TMAs is required to guide effective treatment. Investigators hypothesize that an aHUS-type TMA, related to dysregulation of the alternative complement pathway, is involved and will be characterized by elevated plasma levels of C5b-9 and detectable C5b-9 deposition in bone marrow sinusoidal vessels. Investigators further hypothesize that treatment with inhibitors of terminal complement components will reverse the TMA in vivo, and block endothelial cell damage in our in vitro model systems. The data investigators generate from this observational study of TA-TMAs should enable prediction of their development prior to overt clinical manifestations, and guide appropriate therapy.

DETAILED DESCRIPTION:
Investigators plan to enroll 120 adult patients who are undergoing an allogeneic hematopoietic stem cell transplant and follow them serially for one year. Investigators will harvest and store at -80oC plasma and PBMCs, and collect bone marrow core biopsy specimens on all individuals at baseline, days 28, 100, 190, 365 post-transplant, and at time of relapse of primary disease relapse or TMA development. These time points, bone marrow procedures, and blood draws are part of the ordinary and customary followup of any allogeneic HSCT patient at our institution. With these patient samples investigators will:

1. Determine the incidence of all TMAs fitting the criteria of a Coombs negative hemolytic anemia, thrombocytopenia (25% decrease from baseline) and elevated (2x baseline) LDH, with schistocytes and organ system involvement (typically increased creatinine or new microscopic hematuria or proteinuria)
2. Determine the incidence of an aHUS-like TMA, i.e., a TMA characterized by ADAMTS13 activity in plasma >5% with clinical and laboratory findings which persists after stopping their calcineurin or mTOR inhibitor for one half life (3-7 days, depending on the drug), and ruling out or treating an underlying systemic infection or GvHD.
3. Determine complement component activation, proinflammatory cytokine profile, and baseline complement mutations. This will include ELISA-based measures of plasma C5a, C5b-9, MASP-1-3, tumor necrosis factor(TNF)-α, and interferon-γ, and pre-transplant complement mutational analysis .
4. Assay participants plasma for the ability to induce injury in primary human microvascular endothelial cells (MVEC), and the ability of an anti-C5 monoclonal antibody (mAb) (Alexion, eculizumab (Soliris)) and anti-MASP2 (Omeros, OMS721) mAb, to block these changes in the investigators' established model.
5. Define the degree of C5b-9 deposition in sinusoidal CD34+ endothelial cells by immunohistochemistry, (IHC) examining marrow core biopsies collected at each patient visit and at time of TMA development.
6. Correlate changes in plasma biomarkers, marrow sinusoidal C5b-9 deposition, and the in vitro plasma-MVEC injury model with treatment interventions and treatment outcomes, chosen by the transplant attending of record in this observational cohort.

ELIGIBILITY:
Inclusion Criteria:

* participants scheduled to undergo an allogeneic stem cell transplant
* willing to consent to genetic testing

Exclusion Criteria:

* pregnant women
* nursing mothers
* women of child-bearing potential who are unwilling to use medically accepted methods of contraception
* patients with known contraindications to use of eculizumab
* patients who cannot tolerate plasma exchange

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (age 18-65) undergoing an allogeneic hematopoietic stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with thrombotic microangiopathy occurring in the allogeneic stem cell transplant setting | 2 years
  Per protocol a thrombotic microangiopathy is defined as development of:
  * increase in number of schistocytes per high power microscopic field from baseline
  * increase in baseline level of anemia, measured by hemoglobin decline, which must be Coombs negative
  * unexplained doubling from baseline of serum LDH
Number of participants with allogeneic stem cell transplant-linked TMA persisting after control of infection, GvHD and altering medications | 2 years
  Investigators will determine the number of participants with TMAs that persist after:
  * stopping calcineurin and mTOR inhibitor use for one half-life (3-7 days, depending on drug)
  * treating an underlying infection, if identified
  * suppressing new GvHD, if present

SECONDARY OUTCOMES:
Number of participants with allogeneic stem cell transplant-linked TMA persisting after control of infection, GvHD and altering medications responsive to intervention | 2 years
  This is an observational study. No interventions are specified, by standards of practice could include supportive care, plasma exchange, use of eculizumab (Soliris)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Laurence, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- [Result] Chapin J, Shore T, Forsberg P, Desman G, Van Besien K, Laurence J. Hematopoietic transplant-associated thrombotic microangiopathy: case report and review of diagnosis and treatments. Clin Adv Hematol Oncol. 2014 Sep;12(9):565-73. PMID 25654478